CLINICAL TRIAL: NCT05567276
Title: Non-Violent Resistance Parental Training Versus Treatment as Usual for Children and Adolescents With Severe Tyrannical Behaviour: a Randomized Controlled Trial
Brief Title: Responding to Children and Adolescents With Tyrannical Behaviour
Acronym: REACT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0155
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Oppositional Defiant Disorder
Keywords: Child-To-Parent Violence; Severe tyrannical behaviour; NVR; parental training program
MeSH Terms: conditions — Oppositional Defiant Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group : Non-Violent Resistance parental training (NVR)
  Interventions: Behavioral: Non-Violent Resistance parental training
- Group 2: Group 2 : Treatment as usual (TAU) = Control

INTERVENTIONS:
Behavioral: Non-Violent Resistance parental training — Non-Violent Resistance parental training
  Groups: Group 1

SUMMARY:
This was a randomized controlled trial that compared the NVR intervention group with a TAU group during a four-months period in reducing stress in parents of children aged 6-20 years and displaying severe tyrannical behaviour (STB).

ELIGIBILITY:
Inclusion criteria:

1. being the parent of a child aged 6 - 20 years who endorses the DSM-5 criteria of IODD. In fact, ODD is considered a necessary but not a sufficient condition for tyranny behavior
2. two or more positive answers to the custom quetions routinely used to identify STB in children/adolescents at the University Hospital of Montpellier), related to a 12 month period :

   * Are you afraid of your child?
   * Is your child physically or psychologically violent toward you?
   * Do you think that your child is the decision maker in the family?
   * Do you feel ashamed by your situation at home?
3. being able to attend half of the sessions.

Exclusion criteria:

1. predicted absence from at least half of the sessions
2. subject deprived of liberty
3. subject under guardianship or curatorship.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Parents of children with STB aged 6-20 years old
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Parenting Stress Index/Short Form(PSI-SF) | 4 months from baseline
  Parenting Stress Index/Short Form(PSI-SF) : PSI-SF has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 4 months from baseline
  Hospital Anxiety and Depression Scale (HADS) : HADS is a 14-item measure designed to assess anxiety and depression symptoms in adults. Items are rated on a 4-point severity scale. The HADS produces a scale for anxiety (HADS-A) and for depression (HADS-D). To screen for parental anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores: scores of 7 or less are considered no symptomatology; scores between 8 and 10 are considered doubtful symptomatology; scores of 11 and more are considered definite symptomatology."
Child Behaviour Checklist (CBCL) | 4 months from baseline
  Child Behaviour Checklist (CBCL) : CBCL has 115-item and uses T-scores which allows a wide-ranging evaluation of the child's behavioural profile.
  Raw scores are calculated and used to generate T-scores for eight clinical subscales, two composite scales, one total scale, and four competence scales.
  T-scores ≥70 are in the clinical range for the clinical subscales, T-scores ≥64 are in the clinical range for the composite scales and total scale, and T-scores ≤30 are in the clinical range for the competence scales. Emotional dysregulation was defined as an aggregate T-score of ≥210 on the Attention Problems, Aggressive Behavior, and Anxious/Depressed scales
Strength and Difficulties Questionnaire (SDQ) | 4 months from baseline
  Strength and Difficulties Questionnaire (SDQ) : The SDQ consists of 5 subscales, each containing 5 items. The scales measure emotional symptoms, conduct problems, hyperactivity-inattention, peer relationship problems, and prosocial behaviours.
  Each psychological attribute is scored on a 0-10 scale. A score of 0 is the best outcome concerning the emotional, conduct, hyperactivity, and peer relationship fields (note that these four attributes add up to a total difficulties/overall stress score scored on a 0-40 scale). This scoring reverses for pro-social/score for kind and helpful behaviour, where a score of 10 shows the least amount of difficulty
Kiddie Schedule for Affective Disorders and Schizophrenia Present/Lifetime version | at baseline
  Kiddie Schedule for Affective Disorders and Schizophrenia Present/Lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Diane Purper-Ouakil, M.D., Ph. D., Study Director — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Fongaro E, Aouinti S, Picot MC, Pupier F, Omer H, Franc N, Purper-Ouakil D. Non-violent resistance parental training versus treatment as usual for children and adolescents with severe tyrannical behavior: a randomized controlled trial. Front Psychiatry. 2023 May 4;14:1124028. doi: 10.3389/fpsyt.2023.1124028. eCollection 2023. PMID 37215679